CLINICAL TRIAL: NCT02804022
Title: Vital-signs-integrated Patient-assisted Intravenous Opioid Analgesia for Postsurgical Pain: A Novel Modality to Improve Patient Safety by Detecting and Preventing Respiratory Depression
Brief Title: Vital-signs-integrated Patient-assisted Intravenous Opioid Analgesia
Acronym: VPIAmorphine
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015/3062
Record Dates: First submitted 2016-02-28; First posted 2016-06-17 (Estimated); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Respiratory Depression
Keywords: Respiratory Depression
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VPIA analgesia system (Experimental): Vital-signs-integrated patient-assisted intravenous opioid analgesia system (VPIA). The vital signs (oxygen saturation, respiratory rate, heart rate) will be close monitored when patients is using VPIA pump. The drug used is intravenous morphine (1mg per milligram) with bolus of 1 mg.
  Interventions: Device: VPIA analgesia; Drug: Morphine

INTERVENTIONS:
Device: VPIA analgesia — Recruited subjects will be given a VPIA device containing 1mcg/ml of morphine. Morphine will be administered via an intravenous infusion line with an anti-reflux valve to ensure precise drug administration and no backflow.
  Other Names: VPIA delivery system
Drug: Morphine — Recruited subjects will be given a VPIA device containing 1mcg/ml of morphine. Morphine will be administered via an intravenous infusion line.
  Other Names: Morphine-VPIA

SUMMARY:
This is a closed-loop system which is embodied in a novel and intelligent algorithm that takes into account patients' vital signs. The system allows better and responsive titration of personalized pain relief together with non-invasive physiological monitoring that measures oxygenation, breathing and heart rate continuously.

DETAILED DESCRIPTION:
A glaring safety gap in the administration of commonplace Patient Controlled Analgesia (PCA) opioids unfortunately exists. A significant proportion of patients may suffer from respiratory depression with the use of PCA opioids and it is imperative to discover solutions to improve the safety of PCA opioids, therein improving medication safety, enhancing quality of postoperative care and providing economic cost savings. Currently, no continuous monitoring system that integrates an intelligent decision making response exists.

The investigators primary aim is to develop and commercialise a Vital-signs-integrated (using oxygen saturation, respiratory rate, heart rate) Patient-assisted Intravenous opioid Analgesia (VPIA) that can be integrated into the hospital-wide monitoring systems is capable of making intelligent decision making responses to bridge the PCA safety gap within 12 months.

This VPIA delivery system will be a closed-loop system for safety and efficacy. It will be integrated with continuous vital signs monitoring, and provide appropriate response to breach of safety parameters. It will be part of a larger surveillance system that provides tiered medical and nursing alerts to safety parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-70 years old, female
* Healthy participants who are American Society of Anesthesiologists physical status 1 and 2 (with well controlled medical problems)
* Undergoing elective surgery with the intent of using postoperative PCA with morphine for postoperative analgesia

Exclusion Criteria:

* Allergy to morphine
* With significant respiratory disease and obstructive sleep apnea
* Unwilling to place oxygen saturation monitoring devices during study period
* Unable to comprehend the use of patient controlled analgesia
* Pregnant

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female patients undergoing elective surgery in this institution will be recruited. The study site is specialised in providing healthcare only to women and children in Singapore.
Enrollment: 20 (Actual)
Dates: Start 2016-12-29 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of episodes of breech in safety thresholds | 2 days
  Any episode of oxygen saturation <95%, Heart rate <60 bpm or Respiratory rate <8 breaths/min

SECONDARY OUTCOMES:
Pain scores | 2 or 3 days
  Visual pain score 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Ban L Sng, FANZCA, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sng BL, Tan DJ, Tan CW, Han NR, Sultana R, Sia ATH. A preliminary assessment of vital-signs-integrated patient-assisted intravenous opioid analgesia (VPIA) for postsurgical pain. BMC Anesthesiol. 2020 Jun 8;20(1):145. doi: 10.1186/s12871-020-01060-4. PMID 32513113